CLINICAL TRIAL: NCT01451008
Title: Safety Study of Compression Anastomotic Ring-locking Procedure (CARP) in Patients Undergoing Colonic Resection
Brief Title: Compression Anastomosis Using the Compression Anastomotic Ring-locking Procedure (CARP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Carponovum AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARP-002
Record Dates: First submitted 2011-09-26; First posted 2011-10-13 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Cancer; Polyp
Keywords: Anastomosis; Compression; Colon
MeSH Terms: conditions — Neoplasms; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Compression anastomotic ring-locking procedure (CARP) — The Compression anastomotic ring-locking procedure (CARP) device is based on a set of rings to make a compression anastomosis between the intestinal ends.
  Other Names: The rings are called RapAn

SUMMARY:
The intestinal ends must be rejoined after colonic resection. Conventional methods include sutured and stapled anastomoses, which is associated with 3-6% leakage after colonic surgery. The leakage of an anastomosis can cause serious consequences, such as abdominal infections and/or sepsis. Early detection of anastomotic leakage is the best way to avoid serious abdominal infections. The methods that are used today to detect leaks are unfortunately not very accurate. These methods include monitoring symptoms, temperature, and CRP-levels, and performing abdominal examinations and tomography scans. Because of the difficulties in objectively assessing these parameters, the anastomotic leaks are often diagnosed late. When reoperation is required, a permanent stoma may be made at the level of the sigmoid colon. The CARP system has been developed to achieve a safe anastomosis. The CARP is designed to providing an improved contact surface between the two intestinal ends and the ability to precisely investigate the anastomosis during and after surgery using the catheters of the CARP system. Standardized use of the CARP to anastomose the large intestine may provide significant advantages in the field of colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 - 90 years (male or female)
2. Planned resection due to benign or malign disease in the left colon
3. Cognitive ability to take part in the study and understand the information he/she receives about participating in the study

Exclusion Criteria:

1. Urgent medical condition requiring immediate care
2. Health condition classified as ASA IV
3. Albumin level less than 25 g/l
4. Inflammatory bowel disease (IBD) (ulcerative colitis or Crohn´s disease)
5. Disease that requires more than one anastomosis during the surgical procedure
6. Treatment with cortisone and/or other immunosuppressive medications less than one month before surgery
7. Contraindications to general anaesthesia
8. Cognitive ability that limits the patient's ability to take part in the study and understand the information he/she received about participating in the study, or the patient does not agree to join the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Complications, including anastomotic leakage, problems with ring evacuation | Up to 14 days after operation

SECONDARY OUTCOMES:
Time to evacuation of the CARP device | 1-2 week after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Skåne County, Sweden